CLINICAL TRIAL: NCT04954209
Title: Comparative Study in Long-term Commitment to Physical Activity After Two Different Resumption Programs
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Comité Départemental Olympique et Sportif de Seine Saint Denis (Other)
Responsible Party: Sponsor
Other Study IDs: PERSISTE
Record Dates: First submitted 2021-06-25; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Chronic Disease
Keywords: physical activity
MeSH Terms: conditions — Chronic Disease; Motor Activity | interventions — Exercise; Hospitals

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hospital program of resumption: Program of resumption with physical activities in the hospital
  Interventions: Other: Physical activities in hospital
- Non hospital program of resumption: Program of resumption outside hospital with discovery sessions
  Interventions: Other: Physical activity outside hospital

INTERVENTIONS:
Other: Physical activities in hospital — 3 month in a resumption program of physical activity in hospital
  Groups: Hospital program of resumption
Other: Physical activity outside hospital — 3 month in a resumption program of physical activity outside hospital with discovery sessions
  Groups: Non hospital program of resumption

SUMMARY:
Although physical activity remains an essential pillar of chronicle diseases treatment, long-term adherence to physical activity (PA) continues to prove problematic. A 2019 meta-analysis as well as an overview on the treatment of chronic diseases through physical activity recommend the development of strategies for long-term adherence. Several research paths should be considered in this context.

Through the observation and the comparison of two different programs, the aim of this study is to explore what determining factors will predispose patients to include physical activity in their lifestyle and make a long-term commitment to it/to exercising.

DETAILED DESCRIPTION:
Research design This is a multi-center, longitudinal, minimal risk, category 2 observational comparative study with a convergent parallel mixed method design (Creswell 2015).

The work and intervention arrangements of the two gateway programs are not altered by the research protocol, so the follow-up is strictly observational. As such, it should not affect the usual framework of care and follow-up of patients followed for a long-term condition.

It is a comparative study because it is based on the observation of 2 structures whose methods of care by the PA differ for the same objective.

The patients were followed up during the 3 months of the resumption program and then for 9 months following this program, i.e. 12 consecutive months, which makes it a longitudinal study.

The design is said to be a parallel mixed method study because in the first phase, quantitative data (attendance, quality of life, motivation via questionnaires) and qualitative data (interviews on the reasons for continuing or abandoning PA practice) are collected and analyzed at the same time and analyzed separately. QUANT+QUAL In the second phase, these data are combined in order to integrate the results from the quantitative and qualitative methods, which should allow for a cross-interpretation of the results. Using the convergent parallel mixed method, the qualitative data will complement the quantitative data in order to analyze PA behavior in relation to the interviews on factors that modified PA practice.

Process Data will be collected at T0 inclusion (at enrollment in the resumption program), at 3 months (end of the resumption program), at 6 and 12 months after inclusion.

Inclusion in the study (T0) will be performed by the physical activity educators at the time of enrollment in the corresponding resumption program. The study will be presented to patients meeting the inclusion criteria. And the physical activity educator will inform the patient and collect orally the patient's non-opposition to participate, as well as the non-opposition to the use of the patient's data. If the patient agrees, the physical activity educator will proceed to collect the following data: socio-demographic data, IPAQ, SF-12. The patient will then be informed of a forthcoming physical or telephone appointment for a semi-structured interview with the principal investigator on the reasons for entering the program. The patient will be given a letter of information about the progress of the study with the contact information of the principal investigator.

At the end of enrolment (T0), a copy of the inclusion form, the identification form and the data collected will be sent by email to the principal investigator who will anonymise them.

During 3 months, until T1, the program investigator collects the attendance data of each patient.

At T1, i.e. T0 + 3 months, the corresponding resumption program investigator transmits the attendance data as well as the data from the IPAQ, SF-12 and IMI tests collected during the orientation interview at the end of the program. Patients are informed of a future physical or telephone interview about intra-program factors that have changed PA behavior. Patients are also informed again about the further course of the study (interviews at 6 months and 1 year). In case of absence or temporary impossibility to complete all the tests with the physical activity educator, they can be carried out during a telephone interview.

At T2, i.e. T0 + 6 months, the principal investigator will meet the participants physically or by telephone 6 months (+/- 3 weeks) after their entry into the program. During this interview, the IPAQ, SF-12, and IMI tests were administered, as well as a semi-structured interview on the factors that allowed participants to maintain their PA and their PA practice over the past 3 months.

At T3, i.e., T0 + 12 months, the principal investigator conducted a physical or telephone interview with the participants 12 months (+/- 3 weeks) after they entered the program. During this interview, the IPAQ, SF-12 and IMI tests were administered, as well as a semi-structured interview on the factors allowing the maintenance of PA and the PA practice of the last 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults with a chronic disease
* Consenting
* medical aptitude to physical activity
* registrated in one of the two resumption programs

Exclusion Criteria:

* Doing less than a session of physical activity per week during the resumption program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with a chronic disease who don't practice physical activity, which is part of the treatment
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Practice of physical activity | 12 month
  During a year we follow the physical activity rate with the IPAQ questionary and interviews. With interviews we also question the kind of physical activity.

SECONDARY OUTCOMES:
Self-reported perceptions of quality of life | 12 month
  The evaluation of the quality of life will be measured at 4 points of the study via the SF-12 questionnaire.
  The SF-12 is a general health assessment questionnaire derived from the SF-36: it combines synthetic information with a score on the physical dimension and a score on the mental dimension. It includes 12 items, divided into the same 8 dimensions as the SF-36 (physical activity; life and relationships with others; physical pain; perceived health; vitality; limitations due to psychological state; limitations due to physical state; psychological health. These eight dimensions are used to measure two summary scores of the quality of life of individuals: the physical composite score (PCS) and the mental composite score (MCS) (Leplège Alain, 2001).
  Each quality of life score will be compared with the different phases of physical activity in order to monitor its evolution and influence on adherence to physical activity and its continuation.
Perceptions of enjoyment in practice of physical activity | 12 month
  The enjoyment of physical activity will be measured at three points in the study, T1, T2 and T3, using the Intrinsic Motivation Inventory (IMI) questionnaire (McAuley et al., 1989). This scale determines the pleasure taken in the practice of physical activity over a given period. Using 4 statements (e.g., "I liked the activities I did"), responses are rated on a scale of 1 to 5 from "strongly disagree" to "strongly agree. A high score is synonymous with great pleasure in practicing physical activity.
  Each score will be compared to the different phases of physical activity in order to follow the evolution and the influence of pleasure in the practice for its adherence and continuation.
The qualitative motivational criteria of physical activity practice | 12 month
  The qualitative motivational criteria collected through 4 semi-structured interviews:
  * at T0: reasons for entering the program
  * at T1: intra-program factors that modified PA behavior
  * at T2: information on PA practice following the program: supervised (what type of structure), independent, activity(ies) practiced + factors allowing PA maintenance and PA practice in the last 3 months
  * at T3: information on PA practice following the program: supervised (what type of facility), independent, activity(ies) practiced + factors allowing PA maintenance and PA practice in the last 6 months

OTHER OUTCOMES:
Impact of discovery sessions | 12 month
  With interviews we'd like to know the influence of discovery sessions on the long-term commitment in practice of physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Riquier, PhD std, Principal Investigator — Comité Départemental Olympique et Sportif de Seine Saint Denis / Université de Lorraine

IPD SHARING:
Plan to Share IPD: No
All individual informations will be anonymous

REFERENCES:
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Omorou AY, Langlois J, Lecomte E, Briancon S, Vuillemin A. Cumulative and bidirectional association of physical activity and sedentary behaviour with health-related quality of life in adolescents. Qual Life Res. 2016 May;25(5):1169-78. doi: 10.1007/s11136-015-1172-7. Epub 2015 Nov 6. PMID 26542533
- [Background] Vuillemin A, Boini S, Bertrais S, Tessier S, Oppert JM, Hercberg S, Guillemin F, Briancon S. Leisure time physical activity and health-related quality of life. Prev Med. 2005 Aug;41(2):562-9. doi: 10.1016/j.ypmed.2005.01.006. PMID 15917053
- [Background] Lewis BA, Williams DM, Frayeh A, Marcus BH. Self-efficacy versus perceived enjoyment as predictors of physical activity behaviour. Psychol Health. 2016;31(4):456-69. doi: 10.1080/08870446.2015.1111372. Epub 2015 Nov 18. PMID 26541890
- [Background] Crain AL, Martinson BC, Sherwood NE, O'Connor PJ. The long and winding road to physical activity maintenance. Am J Health Behav. 2010 Nov-Dec;34(6):764-75. doi: 10.5993/ajhb.34.6.11. PMID 20604700
- [Background] Williams NH, Hendry M, France B, Lewis R, Wilkinson C. Effectiveness of exercise-referral schemes to promote physical activity in adults: systematic review. Br J Gen Pract. 2007 Dec;57(545):979-86. doi: 10.3399/096016407782604866. PMID 18252074
- [Background] Gandek B, Ware JE, Aaronson NK, Apolone G, Bjorner JB, Brazier JE, Bullinger M, Kaasa S, Leplege A, Prieto L, Sullivan M. Cross-validation of item selection and scoring for the SF-12 Health Survey in nine countries: results from the IQOLA Project. International Quality of Life Assessment. J Clin Epidemiol. 1998 Nov;51(11):1171-8. doi: 10.1016/s0895-4356(98)00109-7. PMID 9817135
- [Background] McAuley E, Duncan T, Tammen VV. Psychometric properties of the Intrinsic Motivation Inventory in a competitive sport setting: a confirmatory factor analysis. Res Q Exerc Sport. 1989 Mar;60(1):48-58. doi: 10.1080/02701367.1989.10607413. PMID 2489825
- [Derived] Riquier O, Vuillemin A, Van Hoye A. PERSISTE: a mixed methods protocol to identify barriers and levers to a sustainable physical activity practice among patients with chronic disease after physical activity resumption programs. BMJ Open Sport Exerc Med. 2022 Jan 7;8(1):e001261. doi: 10.1136/bmjsem-2021-001261. eCollection 2022. PMID 35070353
- See also: Economic impacts of chronic diseases in France, 2018 — https://drees.solidarites-sante.gouv.fr/sites/default/files/er1077.pdf
- See also: Disparities in the practice of physical activities in France in 2019 — https://www.inegalites.fr/Activites-sportives-des-pratiques-inegales
- See also: Physical activity : treatment of chronic diseases, a collective expertise of INSERM — https://www.inserm.fr/information-en-sante/expertises-collectives/activite-physique-prevention-et-traitement-maladies-chroniques